CLINICAL TRIAL: NCT02001948
Title: The Comparison of Two Different Doses of Morphine Added to Spinal Bupivacaine for Inguinal Hernia Repair.
Brief Title: Intrathecal Morphine for Inguinal Hernia Repair.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Basak Ceyda MECO, MD, DESA, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-02-09
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Inguinal Hernia; Nausea; Vomiting; Pruritus; Postoperative Pain
Keywords: Spinal anaesthesia; morphine; postoperative analgesia; vomiting
MeSH Terms: conditions — Hernia, Inguinal; Nausea; Vomiting; Pruritus; Pain, Postoperative | interventions — Premedication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intrathecal morphine 0.1 mg (Active Comparator): After routine monitorisation, intravenous cannulation and premedication, patients in this group will receive a spinal anaesthesia with 0.1 mg morphine combined with 7.5 mg heavy bupivacaine
  Interventions: Drug: intrathecal morphine 0.1 mg combined with intrathecal heavy bupivacaine 7.5 mg; Device: standard monitoring with Datex Ohmeda anesthesia monitor, GE, Finland; Drug: intravenous cannulation and premedication
- 0.4 mg of intrathecal morphine (Active Comparator): After routine monitorisation, intravenous cannulation and premedication, patients in this group will receive spinal anesthesia with 0.4 mg of morphine combined with 7.5 mg of heavy bupivacaine.
  Interventions: Drug: intrathecal morphine 0.4 mg combined with intrathecal heavy bupivacaine 7.5 mg; Device: standard monitoring with Datex Ohmeda anesthesia monitor, GE, Finland; Drug: intravenous cannulation and premedication

INTERVENTIONS:
Drug: intrathecal morphine 0.1 mg combined with intrathecal heavy bupivacaine 7.5 mg
  Arms: intrathecal morphine 0.1 mg
Drug: intrathecal morphine 0.4 mg combined with intrathecal heavy bupivacaine 7.5 mg
  Arms: 0.4 mg of intrathecal morphine
Device: standard monitoring with Datex Ohmeda anesthesia monitor, GE, Finland — electrocardiography, heart rate, pulse oximetry and noninvasive arterial blood pressure
Drug: intravenous cannulation and premedication — 18-gauge intravenous cannula was inserted at the forearm opposite to the surgical side and routine iv premedication (midazolam 0.03 mg/kg) was given

SUMMARY:
The aim of this study was to compare the effects of two different doses of intrathecal morphine (0.1 mg and 0.4 mg) combined with 7.5 mg of heavy bupivacaine on postoperative block regression times, postoperative analgesia and the severity of side effects, for inguinal hernia repairs.

DETAILED DESCRIPTION:
The purpose of this study was to compare spinal anesthesia with low dose heavy bupivacaine combined with 0.1 mg or 0.4 mg of morphine in inguinal hernia repair surgeries. Anesthesia onset time (sensory and motor blocks) as well as postoperative recovery (first mobilisation, first voiding) time were compared. Also the postoperative pain management and side effects (nausea, vomiting and pruritus) were assessed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology physical status I-II patients
* aged 18-65 years
* undergoing elective unilateral open inguinal hernia repair surgery

Exclusion Criteria:

* contraindications to spinal anesthesia
* central or peripheral neuropathies
* severe respiratory or cardiac diseases
* chronic analgesic use
* history of substance abuse
* allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sensory and motor block | The change in motor block and sensory block levels will be assessed after performing spinal block, every 5 minutes for 30 minutes and then at the end of the procedure.
  Sensory and motor block produced by the spinal anaesthesia will be assessed prior the procedure to define readiness for surgery and then once the procedure is over, sensory and motor block levels will be assessed one more time to follow up the block regression times. Motor block will be assessed with Bromage scale (0: no motor block, 1: hip blocked; 2: hip and knee blocked; 3: hip, knee and ankle blocked). Sensory block will be assessed using loss of pinprick sensation. The onset of surgical anesthesia is defined as loss of pinprick sensation at ≥ T10 with a Bromage score ≥ 2.

SECONDARY OUTCOMES:
first mobilisation, first urination and first analgesic times | after the procedure, during the first 24 hours
  all patients will be followed up during the first postoperative 24 hours to assess the first mobilisation, first voiding and first analgesic requirement times.

OTHER OUTCOMES:
postoperative nausea, vomiting and pruritus | after the procedure, during the first 24 hours
  All patients will be followed up for the first postoperative 24 hours to determine the nausea, vomiting and pruritus incidences.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Ceyda Meco, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Ibni Sina Hospital general surgery OR, Ankara, Turkey (Türkiye)